CLINICAL TRIAL: NCT02027935
Title: Phase II Study of Cellular Adoptive Immunotherapy Using Autologous CD8+ Antigen-Specific T Cells and Anti-CTLA4 for Patients With Metastatic Melanoma
Brief Title: CD8+ Antigen-Specific T Cells, Cyclophosphamide, Aldesleukin, and Ipilimumab in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-1055; NCI-2014-01040 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-1055 (Other: M D Anderson Cancer Center); P50CA159981 (NIH)
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Melanoma; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Cyclophosphamide; Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (T cells, chemo, aldesleukin, ipilimumab) (Experimental): Beginning 48 to 72 hours prior to T cell infusion, patients receive cyclophosphamide IV over 30-60 minutes. Patients then receive autologous CD8+ melanoma-specific T cells IV over 30-60 minutes on day 0, aldesleukin SC BID on days 0-13 and ipilimumab IV over 90 minutes on days 1, 22, 43, and 64 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Aldesleukin; Biological: Autologous CD8+ Melanoma Specific T Cells; Drug: Cyclophosphamide; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Autologous CD8+ Melanoma Specific T Cells — Given IV
  Other Names: Autologous Melanoma Specific Cytotoxic T Lymphocytes
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well white blood cells taken from person's own (autologous) cluster of differentiation (CD)8+ antigen-specific T cells, cyclophosphamide, aldesleukin, and ipilimumab work in treating patients with melanoma that has spread to another place in the body. Autologous CD8+ antigen-specific T cells are white blood cells that are designed in the laboratory to find melanoma cells and may kill them. Biological therapies, such as aldesleukin, use substances made from living organisms that may stimulate the immune system in different ways and stop tumor cells from growing. Immunotherapy with monoclonal antibodies, such as ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving autologous CD8+ antigen-specific T cells with cyclophosphamide, aldesleukin, and ipilimumab may be an effective treatment for patients with metastatic melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the safety and efficacy of adoptively transferred cytotoxic T-lymphocytes (CTL) targeting melanoma tumors combined with anti-CTLA4.

SECONDARY OBJECTIVES:

I. Evaluate the influence of anti-CTLA4 on the duration of in vivo persistence and anti-tumor efficacy achieved following adoptive transfer of antigen-specific CTL.

II. Evaluate the influence of anti-CTLA4 on the induction of T cells to non-targeted tumor-associated antigens (antigen-spreading) following adoptive transfer antigen-specific CTL, and the correlation of these responses with clinical outcome.

OUTLINE:

Beginning 48 to 72 hours prior to T cell infusion, patients receive cyclophosphamide intravenously (IV) over 30-60 minutes. Patients then receive autologous CD8+ melanoma-specific T cells IV over 30-60 minutes on day 0, aldesleukin subcutaneously (SC) twice daily (BID) on days 0-13 and ipilimumab IV over 90 minutes on days 1, 22, 43, and 64 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY FOR ENROLLMENT
* Histopathologic documentation of melanoma concurrent with the diagnosis of metastatic disease
* Expression of human leukocyte antigen (HLA)-A2
* Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status of '0-1' at screening visit
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized; suggested precautions should be used to minimize the risk of pregnancy for at least 1 month before start of therapy, and while women are on study for up to 3 months after T cell infusion, and at least 8 weeks after the study drug is stopped; WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal
* Men must be willing and able to use an acceptable method of birth control, for at least 3 months after completion of the study, if their sexual partners are WOCBP
* Willing and able to give informed consent
* Adequate venous access - consider peripherally inserted central catheter (PICC) or central line
* Evaluation of v-raf murine sarcoma viral oncogene homolog B (BRAF)V600 mutation status
* Measurable tumor (by Response Evaluation Criteria in Solid Tumors [RECIST] criteria)
* Melan-A (MART) 1 or solute carrier family 45, member 2 (SLC45A2) (+) staining results; (if patients have not had staining test in the past, the test will be run after patient consent is obtained, but before enrollment)
* ELIGIBILITY FOR TREATMENT (INCLUDES CYCLOPHOSPHAMIDE, T CELL, ANTI-CTLA4 INFUSIONS AND SC IL-2)
* ECOG/Zubrod performance status of '0-1'
* At least 4 weeks must have elapsed since the last chemotherapy, radiotherapy or major surgery; at least 6 weeks for nitrosoureas, mitomycin C and liposomal doxorubicin; if started before T-cell administration, ipilimumab infusions must be least 21 days apart
* Toxicity related to prior therapy must either have returned to =< grade 1, baseline, or been deemed irreversible
* Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 8 weeks after study drug is stopped
* Willing and able to give informed consent.

Exclusion Criteria:

* EXCLUSION FOR ENROLLMENT
* Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix
* Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception; women of childbearing potential with a positive pregnancy test within 3 days prior to entry
* Active and untreated central nervous system (CNS) metastasis (including metastasis identified during screening magnetic resonance imaging [MRI] or contrast computed tomography [CT])
* No signs or symptoms of CNS metastases (mets) within the last 30 days (from enrollment evaluation)
* No single lesion larger than 1 cm
* No more than 5 lesions
* Autoimmune disease: patients with a history of inflammatory bowel disease are excluded from this study, as are patients with a history of autoimmune disease (e.g. systemic lupus erythematosus, vasculitis, infiltrating lung disease) whose possible progression during treatment would be considered by the investigator to be unacceptable
* Any underlying medical or psychiatric condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea
* Positive screening tests for human immunodeficiency virus (HIV), hepatitis B (hep B), and hepatitis C (hep C) (referencing blood draw at leukapheresis screening); if positive results are not indicative of true active or chronic infection, the patient can be treated
* White blood cells (WBC) =< 1000/uL
* Hematocrit (Hct) =< 24% or hemoglobin (Hb) =< 8 g/dL
* Absolute neutrophil count (ANC) =< 500
* Platelets =< 50,000
* Creatinine >= 3.0 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >= 2.5 x ULN
* Bilirubin >= 3 x ULN
* Steroids are not permitted 3 days prior to T cell infusion and concurrently during therapy
* Any non-oncology vaccine therapy used for the prevention of infectious disease within 1 month before or after any ipilimumab dose
* Patients may not be on any other treatments for their cancer aside from those included in the protocol; patients may not undergo another form of treatment concurrently with this study
* EXCLUSION CRITERIA FOR TREATMENT
* WBC =< 1000/uL (prior to cyclophosphamide and T cell infusions)
* Hct =< 24% or hemoglobin =< 8 g/dL (prior to cyclophosphamide and T cell infusions)
* ANC =< 500 (prior to cyclophosphamide and T cell infusions)
* Platelets =< 50,000 (prior to cyclophosphamide and T cell infusions)
* Creatinine >= 3.0 x ULN (prior to cyclophosphamide and T cell infusions)
* AST/ALT >= 2.5 x ULN (prior to cyclophosphamide and T cell infusions)
* Bilirubin >= 3 x ULN (prior to cyclophosphamide and T cell infusions)
* Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception; women of childbearing potential with a positive pregnancy test within 3 days prior to entry.
* Steroids are not permitted 3 days prior to T cell infusion and concurrently during therapy.
* Any non-oncology vaccine therapy used for the prevention of infectious disease within 1 month before or after any ipilimumab dose.
* Patients may not be on any other treatments for their cancer aside from those included in the protocol. Patients may not undergo another form of treatment concurrently with this study.
* Active and untreated central nervous system (CNS) metastasis (including metastasis identified during screening MRI or contrast CT):

  * No signs or symptoms of CNS mets within the last 30 days (from enrollment evaluation).
  * No single lesion larger than 1cm
  * No more than 5 lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adi Diab, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Phase II trial aimed at treating up to 20 HLA-A*0201+ individuals with metastatic melanoma. A perfomance status of >70% (85% of total patients, n-119) and HLA-A@ expression (40% of these patients), an average of 45 patients/year will be eligible for this study
Pre-assignment Details: 16 subjects consented; 7 subjects treated
Groups:
- Treatment (T Cells, Chemo, Aldesleukin, Ipilimumab): Single dose of cytoxan at 300mg/m2 on Day-2; Day 0 infusion of 10^10 T cells/2; 14-day course of low-dose s.c. IL-2; Anti-CTLA4 3 mg/kg IV over 90 minutes 24 hrs post T Cell infusion; Anti-CTLA4 q3 weeks 3 mg/kg IV for 4 doses.
Period: Overall Study
Arm/Group | Treatment (T Cells, Chemo, Aldesleukin, Ipilimumab)
Started | 7
Completed | 0
Not Completed | 7
Not completed — Death | 1
Not completed — Lack of Efficacy | 5
Not completed — Study Closure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (T Cells, Chemo, Aldesleukin, Ipilimumab)
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: CTL With Anti-CTLA4
Description: Evaluate the safety and efficacy of adoptively transferred CTL targeting melanoma tumors combined with anti-CTLA4
Time Frame: Baseline up to 2 years
Population: Data was not collected
Arm/Group | Treatment (T Cells, Chemo, Aldesleukin, Ipilimumab)
Number analyzed (Participants) | 0

2. Secondary Outcome: Anti-CTLA4 Duration
Description: Evaluate the influence of anti-CTLA4 on the duration of in vivo persistence and anti-tumor efficacy achieved following adooptive transfer of antigen-specific CTL.
Time Frame: Baseline up to 2 years
Population: Data was not collected
Arm/Group | Treatment (T Cells, Chemo, Aldesleukin, Ipilimumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 2 years
Description: CTCAE v4.0
Arm/Group | Treatment (T Cells, Chemo, Aldesleukin, Ipilimumab)
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 7/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (T Cells, Chemo, Aldesleukin, Ipilimumab) (N=7)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hyponatremia (Investigations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hypotention (Cardiac disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Lymphedema (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (T Cells, Chemo, Aldesleukin, Ipilimumab) (N=7)
Creatinine increased (Investigations) | 3 (4)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (8)
Dizziness (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Endocrine disorders (Endocrine disorders) | 1 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Eye disorders (Eye disorders) | 2 (3)
Eye pain (Eye disorders) | 1 (1)
Fatigue (General disorders) | 4 (14)
Fever (General disorders) | 3 (10)
Gait disturbance (General disorders) | 1 (1)
Gastrointestinal disordedrs (Gastrointestinal disorders) | 2 (3)
General disorders (General disorders) | 3 (5)
Headache (Nervous system disorders) | 5 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot Flashes (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (7)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypothyrodism (Vascular disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Lymphedema (Vascular disorders) | 2 (4)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness lower limbs (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 6 (7)
Non-cardiac chest pain (Cardiac disorders) | 1 (2)
Pain (Gastrointestinal disorders) | 4 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Psychiatric disorders (Psychiatric disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Watery Eyes (Eye disorders) | 1 (1)
Weight Loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT02027935/Prot_SAP_000.pdf